CLINICAL TRIAL: NCT03845530
Title: The Inflammatory Burden in Hemodialysis vs. Peritoneal Dialysis Patients: the Role of Alpha-defensin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYMC-123-18
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Kidney Failure; Inflammation
MeSH Terms: conditions — Renal Insufficiency; Inflammation | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis group (Active Comparator): Blood sample taken and sent to laboratory for analysis
  Interventions: Diagnostic Test: Blood Test
- Peritoneal dialysis (Active Comparator): Blood sample taken and sent to laboratory for analysis
  Interventions: Diagnostic Test: Blood Test

INTERVENTIONS:
Diagnostic Test: Blood Test — Blood test taken and sent for laboratory analysis

SUMMARY:
The aim of this study is to determine the levels of alpha-defensin throughout the hemodialysis course compared to the levels at the end of a course of peritoneal dialysis, as a reflection of the inflammatory burden.

ELIGIBILITY:
Inclusion Criteria:

* Kidney failure patients undergoing hemodialysis or peritoneal dialysis

Exclusion Criteria:

* Active inflammatory or infectious disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Alpha-Defensin Levels | One year
  Alpha-defensin levels will be compared between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Rami Abu Fanne, MD, PhD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No